CLINICAL TRIAL: NCT04873843
Title: The Impact of Multi-Touch Functional Digital Game on Intelligence and Vitality for the Community-dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-03-011
Record Dates: First submitted 2021-04-05; First posted 2021-05-05 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2021-04

CONDITIONS: Aging
Keywords: Elderly; Functional Digital Game; Multi-touch Game; Intelligence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional digital game training group (Experimental): These functional digital game programs have been developed to improve the intelligence and vitality in the community-dwelling elderly. The program includes sub-categories such as attention, working memory, memory and executive functions with various levels of difficulty.
  Interventions: Behavioral: Functional digital game training group
- Individual cognitive training (Experimental): Individual cognitive training has been used to improve the intelligence and cognitive function in community-dwelling elderly. The program includes sub-categories such as attention, working memory, memory and executive functions with various levels of difficulty.
  Interventions: Behavioral: Individual cognitive training

INTERVENTIONS:
Behavioral: Functional digital game training group — Functional digital game training group is divided in 16 participants. In one session, participants in the functional digital game training group completed 40 minutes of intervention using various functional digital game such as working memory, memory, and attention. (Total 10 session)
  Arms: Functional digital game training group
Behavioral: Individual cognitive training — Functional digital game training group is divided in 16 participants. In one session, participants in the individual cognitive training group completed 40 minutes of intervention using various cognitive training such as working memory, memory, and attention. (Total 10 session)
  Arms: Individual cognitive training

SUMMARY:
This single-blinded, randomized, controlled trial includes 32 elderly. The participants were randomized to intervention(Happy Table) and control(cognitive stimulation activity) groups. Each group is divided in 16 participants. In one session, participants in the Happy Table group completed 40 minutes of intervention using Happy Table serious game, whereas those in the Control group completed 40 minutes of cognitive stimulation game.

DETAILED DESCRIPTION:
At the first visit, the subjects are fully informed of the study if appropriate after determining whether they meet the selection criteria. This single-blinded, randomized, controlled trial includes 32 elderly. The participants were randomized to intervention(Happy Table) and control(cognitive stimulation activity) groups. Each group is divided in 16 participants. In one session, participants in the Happy Table group completed 40 minutes of intervention using Happy Table serious game, whereas those in the Control group completed 40 minutes of cognitive stimulation game.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling senior citizens aged 65 to 84
* Those without a history of central nervous system(CNS) disease

Exclusion Criteria:

* When it is difficult to understand the task performance due to severe cognitive decline(Korean Simple Mental State Test, K-MMSE 10 points or less).
* When it is difficult to use this game device due to problems such as decreased vision or fracture of the upper limb
* In case of accompanying serious mental illness

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance on Stroop test (Neuropsychological test) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  It measures a participant's processing speed, selective attention and inhibitory control. The participant will be asked to read 'word' of the colored words or 'name of the color' of the colored words in separate trials. The main scores produced in this test are completion time and errors. The contrast score of the two trial's completion time means interference.

SECONDARY OUTCOMES:
Change from baseline performance on Fluency Test (Neuropsychological test) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  This is a generative naming test. That measure how many words you can spontaneously speak within a limited time of words that fall into a specific category (e.g. animals, store goods, vegetables) or words starting with a letter (e.g. F • A • S or C·F·L).
Change from baseline performance on Trail Making Test (Neuropsychological test) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  It consists of type A and type B trials. The participant should connect the numbers (1~25) as quickly as possible in Type A trial, and connect the numbers (1~13) and alphabets (A~L) alternatively as quickly as possible in type B trial. The main scores produced in this test are completion time and errors. Higher score means worse performance.
Change from baseline performance on Digit Span Test (Neuropsychological test) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  It measures auditory attention span and includes forward and backward trials. The participant listens to a series of numbers and calls the sequence correctly. The sequence increases in each trial. The final score is the longest number of sequential digits that the participant can remember correctly. The scores range from 3 to 8. The higher the score, the better the performance.
Change from baseline performance on Auditory Verbal Learning test (Neuropsychological test) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  It measures participant's verbal memory. The participant will hear 15 words and recall them immediately and after 20 minutes again. The main scores produced in this test are the numbers of recalled words of the immediate and delayed trials. Immediate memory score is the sum of 5 trial's correct response and score ranges between 0 and 60. Delayed memory score is the correct response of the delayed trial and the score range is 0 to 15. Higher score means better performance.
Change from baseline activity on functional Near-Infrared Spectroscopy (fNIRS) during the intervention(Day 1 and 12)and after intervention completion(Day 12) | Baseline, during the intervention(Day 1 and 12), Through intervention completion(Day 12)
  It measures brain activity during cognitive tasks to see if cognitive training affects brain function.
Change from baseline activity on Contrasting Program/Go-No-Go test after the intervention (Day 13). | Baseline, Day 13(After the intervention)
  The Contrasting Program and go-no go test requires a subject to emit a simple motor response to one cue while inhibiting the response in the presence of another cue. This test has been effective in demonstrating impulsivity (elevated commission error rate) in elderly with attention deficit.
Change from baseline activity on Geriatric Depression Scale (GDS) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  GDS is a 15-item self-report assessment used to identify depression in the elderly. A score of 0 to 5 is normal. A score greater than 5 suggests depression
Change from baseline activity on health-related quality of life instrument with 20 items (HINT-20) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  The total score of the HINT-20 is converted to a 0-100 scale, with higher scores indicating better health-related quality of life.
Change from baseline activity on General Self-Efficacy Scale (GSE) after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  General self-efficacy (GSE), individuals'belief in their ability to perform well in a variety of situations. General self-efficacy (GSE) is the belief in one's competence to attempt difficult or novel tasks, and to cope with adversity arising from specific demanding situations.
Change from baseline activity on International Physical Activity Questionnaire after the intervention (Day 13). | Baseline, After the intervention (Day 13)
  Physical Activity Questionnaire collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour, comprising 16 questions.
User Satisfaction Questionnaire after intervention. | After the intervention (Day 13)
  We evaluate the satisfaction questionnaire for each training.
Change from baseline activity on smart band activity through intervention completion(Day 12). | Baseline, through intervention completion(Day 12)
  Each participant was given an smart band(number of steps count) and instructed to wear it on the wrist during waking hours until completion of the training program. This included both intervening training days (totaling 10).

CONTACTS AND LOCATIONS:
Overall Officials: Yun-hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea